CLINICAL TRIAL: NCT04357522
Title: A Single-center, Randomised, Blind, Similar Vaccine Control, Non-inferior Designed Phase III Clinical Trial to Evaluate Immunogenicity and Safety Study of 15-Valent Pneumococcal Conjugate Vaccine in 2-month-old and 3-month-old Healthy Volunteers
Brief Title: Immunogenicity and Safety Study of 15-Valent Pneumococcal Conjugate Vaccine in 2-month-old and 3-month-old Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201904002
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Received Vaccine: 15-valent pneumococcal Conjugate Vaccine(experimental vaccine), 0.5 ml/dose
  Interventions: Biological: 15-Valent Pneumococcal Conjugate Vaccine
- Positive control group (Active Comparator): Received Vaccine: 13-valent pneumococcal Conjugate Vaccine(positive control vaccine), 0.5 ml/dose
  Interventions: Biological: 13-Valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 15-Valent Pneumococcal Conjugate Vaccine — 4/1 dose(s) according to age of subjects. Single intramuscular dose contains 0.5ml 15-Valent Pneumococcal Conjugate Vaccine.
  Arms: experimental group
Biological: 13-Valent Pneumococcal Conjugate Vaccine — 4/1 dose(s) according to age of subjects. Single intramuscular dose contains 0.5ml 15-Valent Pneumococcal Conjugate Vaccine.
  Arms: Positive control group

SUMMARY:
The purpose of this study is to evaluate Immunogenicity and safety of 15-Valent Pneumococcal Conjugate Vaccine in healthy volunteers aged 2 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 2 months (minimum to 6 weeks), term (37-42 weeks gestation) and birth weight ≥2.5 kg.
* The guardian understands the vaccination and research procedures, volunteers to participate in the research and sign the informed consent.
* The guardian can follow the clinical research program, will be able to follow up until 3 years after booster immunization and have the ability to use thermometers, scale and fill in diary and contact cards as required.
* There was no history of other live vaccines in the past 14 days and no history of other inactivated vaccines in the seventh day.
* Subaxillary body temperature <=37.0 C.
* Determine health based on medical history, physical examination, and researcher's judgment.

Exclusion Criteria:

* Have been vaccinated a listed or experimental pneumococcal vaccine.
* History of invasive diseases caused by Streptococcus pneumoniae confirmed by bacterial culture in the past.
* In the past, there was any history of vaccination or serious allergy to drugs. In the past, fever of over 39.5 C related to vaccination occurred in biological products for vaccination and prophylaxis.
* History of convulsion, epilepsy, encephalopathy and psychiatry or family history.
* Had abnormal labor (dystocia, device midwifery), history of asphyxia rescue and nerve organ damage.
* History of pathological jaundice confirmed by diagnosis.
* A history of thrombocytopenia or other coagulation disorders with definite diagnosis.
* Human serum gamma globulin injection after birth.
* There are known or suspected immunological abnormalities, including immunosuppressive therapy (radiotherapy, chemotherapy, corticosteroids, antimetabolites, cytotoxic drugs), HIV infection, etc.
* Congenital malformations, severe malnutrition, developmental disorders, genetic defects (e.g. broad bean disease).
* Severe chronic disease, infectious disease, active infection, liver disease, kidney disease, cardiovascular disease, malignant tumor.
* Severe asthma.
* Systemic rash, dermatophytes, skin pus or blister.
* Participation in other drug clinical trials.
* Anything that the researcher considers likely to affect the evaluation of the study.

Ages: 6 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1950 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity study endpoint | 30 day after each vaccination
  Percentage of participants with seroresponse to each vaccination
Safety study endpoint | 30 day after each vaccination
  Occurrence of adverse events during a 30 day follow-up period after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Du Lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (3):
- China (3):
  - Daming Center for Disease Control and Prevention, Daming, Hebei
  - Laishui Center for Disease Control and Prevention, Laishui, Hebei
  - Zhengding Center for Disease Control and Prevention, Zhengding, Hebei